CLINICAL TRIAL: NCT04015765
Title: Hybrid-APC Margin Ablation to Prevent Post EMR Adenoma Recurrence
Acronym: h-APC_EMR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Penn State University (Other); University of Milan (Other); Erbe Elektromedizin GmbH (Industry); Unity Health Toronto (Other); University of British Columbia (Other)
Responsible Party: Principal Investigator, Daniel Von Renteln, Principal Investigator, Centre hospitalier de l'Université de Montréal (CHUM)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CE.19.119
Record Dates: First submitted 2019-07-04; First posted 2019-07-11 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Colorectal Cancer; Polyp of Colon
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Polyps

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Group treatment h-APC and EMR (Experimental): Standard endoscopic mucosal resection (EMR) technique will be used for primary removal of all polyps. Submucosal injection will be used to lift the polyp from the muscularis propria. Injection is used as per the current standard of care using a contrast agent and a lifting agent (e.g. NaCl 0.9% or Voluven). Snare electrocautery resection will be facilitated until complete visible removal of the complete polyp. Electrocautery snare technique is facilitated using standard microprocessor controlled electrocautery (e.g. ERBE VIO Endocut 3-1-6). Ablation of the margin after visibly complete removal of the polyp is routinely applied. For thermal ablation hybrid APC (Erbe Hybrid APC) will be applied using standard settings on the margin and resection base. Once resection and thermal ablation is considered complete the mucosal defect can be closed with clips or another preventative measure applied to reduce the risk for post-polypectomy bleeding.
  Interventions: Procedure: Hybrid Argon Plasma Coagulation and EMR procedure

INTERVENTIONS:
Procedure: Hybrid Argon Plasma Coagulation and EMR procedure — Hybrid Argon Plasma Coagulation (h-APC) combines an ablation technique (APC) with the option for submucosal saline injection using a high-pressure water jet. The technique allows to lift dysplastic epithelium thus creating a safety cushion under the mucosa is lifted with a saline injection and then to ablate larger areas more thoroughly and with a higher energy setting, with a low risk for side effects or complications

SUMMARY:
Endoscopic Mucosal Resection (EMR) is the current standard for effective endoscopic resection of such colon adenomas. If resection is possible in one piece (so-called "en bloc" resection) then recurrence rates are low. However, most non-pedunculated polyps >2 cm are removed in pieces ("piece-meal" resection) which leads to disease recurrence rates between 12-30%. In the March 2019 issue of Gastroenterology Bourke et al. presented that post-EMR ablation of the resection margins using soft coagulation with the tip of a resection snare reduces adenoma recurrence to 5% compared to 21% recurrence found in the control group. Hybrid Argon Plasma Coagulation (h-APC) combines an ablation technique (APC) with the option for submucosal saline injection using a high-pressure water jet. The technique allows to lift of dysplastic epithelium thus creating a safety cushion under the mucosa is lifted with a saline injection and then to ablate larger areas more thoroughly and with a higher energy setting, with a low risk for side effects or complications.

The study hypothesis is that routine use of hybrid Argon Plasma Coagulation (h-APC) for ablation of the post-EMR resection margins and resection surface area will reduce post-EMR adenoma recurrence to 5% or lower.

DETAILED DESCRIPTION:
This is a prospective, multi-center study enrolling patients with non-pedunculated colorectal polyps ≥ 20mm for endoscopic mucosal resection (EMR). All primary EMR procedures will combine EMR with h-APC ablation of the base and margins after complete EMR resection to prevent adenoma recurrence.

Schedule of activities

1. Enrollment visit before the endoscopy (ALL PATIENTS), in the outpatient clinic, or before the EMR.

   Eligible patients who have consented to participate in the study will be asked to take a standard colonoscopy preparation before their scheduled procedure.
2. EMR intervention (ALL PATIENTS meeting eligibility criteria). Only if a polyp meets inclusion criteria, the study subject will be enrolled. The standard endoscopic mucosal resection (EMR) technique will be used for the primary removal of all polyps. Submucosal injection will be used to lift the polyp from the muscularis propria. Injection is used as per the current standard of care using a contrast agent and a lifting agent (e.g., NaCl 0.9% or Voluven). Snare electrocautery resection will be facilitated until complete visible removal of the complete polyp. Electrocautery snare technique is facilitated using standard microprocessor-controlled electrocautery. If residual polyp tissue cannot remove by a snare, other means such as cold snare (i.e., for small residual polyp tissue that cannot be engaged into standard snares), hot avulsion technique or Argon plasma coagulation or soft coagulation by the tip of snare can be used.

   The polyp site will be marked with submucosal injection of approximately 1-2cc of India ink (standard of care to mark lesions in the colon safely) to allow recognition at follow-up endoscopy. Polyps are sent to the pathology lab and evaluated according to standard practice by institutional pathologists.19 To determine the homogeneity and depth of h-APC margin ablation in the pathology lab, some ablated margins might be resected using the standard cold snare technique.

   Telephone calls or visits 14-30 days following the EMR will be conducted to assess possible adverse events.
3. Follow-up 1 (FU1, ALL PATIENTS): colonoscopy 4 months (± 2 months) after the EMR intervention with the assessment of the primary outcome (biopsy/pathology-confirmed recurrence at post-EMR site). Patients with visible recurrence at the EMR site will undergo additional h-APC treatment for complete eradication at the first follow-up.
4. Follow-up 2 (ONLY FOR PATIENTS with visible recurrence and biopsy confirmed recurrence at FU1 will undergo FU2 scheduled 4 months (± 2 months) after FU1 (within 1 year after EMR procedure) with the assessment of recurrence/complete eradication rates (biopsy/pathology confirmed complete eradication post-EMR and h-APC at FU1).
5. Patients with not visible but pathology-confirmed recurrence will be rescheduled for another colonoscopy with h-APC treatment of the post-EMR site and another follow-up colonoscopy for biopsies and confirmation of complete/incomplete eradication within 1 year after the initial EMR.

ELIGIBILITY:
Inclusion Criteria:

* All Ethnicity and race
* Patient referred for endoscopic resection of all colorectal polyps non-pedunculated equal or greater 20 mm
* Written informed consent

Exclusion Criteria:

* Patients with known (biopsy proven) invasive carcinoma in a potential study polyp
* Previous partial EMR
* Pedunculated polyps (as defined by Paris Classification type Ip or Isp)
* Patients with ulcerated depressed lesions (as defined by Paris Classification type III)
* Patients with inflammatory bowel disease
* Patients who are receiving an emergency colonoscopy
* Poor general health (ASA class>3)
* Patients with coagulopathy with an elevated INR ≥1.5, or platelets <50
* Poor bowel preparation (Boston bowel prep score ≤2)
* Target sign or perforation during initial EMR
* Need for ESD for complete resection prior to APC
* Pregnancy and breast-feeding.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 376 (Actual)
Dates: Start 2019-08-26 (Actual); Primary Completion 2024-12-13 (Actual); Study Completion 2025-01-08 (Actual)

PRIMARY OUTCOMES:
Post-EMR recurrence at FU1 | 4 months (+- 2 months) after the index h-APC and EMR procedure
  The post-EMR recurrence at FU1 is defined as the rate of first follow-up colonoscopies with found adenomas.

SECONDARY OUTCOMES:
Complete adenoma eradication rates | Within 1 year after the index EMR
  The complete adenoma eradication rate is defined as the rate of follow-up colonoscopies without any adenoma detected within 1 year after the index EMR, with potential re-ablation at FU1 for patients with visible or non-visible, but pathology confirmed adenoma recurrence.
Incidence of complications | 14 days after the index EMR
  The rate of complications including bleeding, perforation, post polypectomy syndrome, and clinical events that require admission to the hospital.
Severe bleeding complication rate | 14 days after the index EMR
  Rate of severe bleeding cases at the time of EMR resection, or during 14 days of follow-up. Immediate severe bleeding is defined as the inability to stop bleeding during the EMR procedure and the need for a non-endoscopic intervention (e.g., surgery or interventional radiology). Delayed severe bleeding is defined as the need for hospitalization, transfusion, a repeat colonoscopy or sigmoidoscopy, surgery, or interventional radiology.
Perforation rate | 14 days after the index EMR
  Rate of colonoscopies with perforation, defined as a complete hole or full-thickness resection of the muscularis propria (Sidney Classification of Deep Mural Injury Type IV).
Post-polypectomy syndrome incidence | 14 days after the index EMR
  Incidence rate of post-polypectomy syndrome, defined as abdominal pain severe enough to warrant an ED visit or hospital admission and presence of leukocytosis and/or required treatment with antibiotics.
Completeness of polyp resection | 14 days after the index EMR
  Number of cases with completeness of thermal ablation of polyp resection margin, defined as the proportion of margins with at least one region of unablated margin as determined by histopathological evaluation of resected ablated margins.
Intraprocedural bleeding rate | During the procedures
  Rate of colonoscopies with immediate bleeding that requires endoscopic intervention to stop the bleeding (e.g., clip placement or soft snare coagulation).
Need for colon resection rate | Within 1 year after the index EMR
  Rate of patients who require surgery for polyp removal or as a result of complications related to the EMR or follow-up procedures.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel von Renteln, MD, PhD, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre Hospitalier Universitaire de Montréal (CHUM), Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures and appendices).
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Beginning 12 months and ending 36 months following article publication.
Access Criteria: Proposals should be directed to daniel.von.renteln.med@ssss.gouv.qc.ca . To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Derived] Motchum L, Levenick JM, Djinbachian R, Moyer MT, Bouchard S, Taghiakbari M, Repici A, Deslandres E, von Renteln D. EMR combined with hybrid argon plasma coagulation to prevent recurrence of large nonpedunculated colorectal polyps (with videos). Gastrointest Endosc. 2022 Nov;96(5):840-848.e2. doi: 10.1016/j.gie.2022.06.018. Epub 2022 Jun 18. PMID 35724695